CLINICAL TRIAL: NCT03165851
Title: Efficacy Analysis of Comparison of CAMS-2005 Trial and CAMS-2009 Trial for Pediatric Acute Myeloid Leukemia
Brief Title: Efficacy Analysis of Comparison of CAMS（Chinese Academy of Medical Sciences）-2005 Trial and CAMS-2009 Trial for Pediatric Acute Myeloid Leukemia
Status: Completed | Type: Observational
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Other Study IDs: RE2016001
Record Dates: First submitted 2017-05-16; First posted 2017-05-24 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2017-05

CONDITIONS: Acute Myeloid Leukemia, Pediatric
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CAMS-2005 trial: The induction course was Daunorubicin(DNR) + Cytarabine(Ara-C) or Homoharringtonine(HHT) + Ara-C or HHT + DNR + Ara-C. There are 5 consolidation course after complete remission (CR).
- CAMS-2009 trial: The induction course was MAE(Mitoxantrone + Cytarabine + Etoposide) or IAE(Idamycin + Cytarabine + Etoposide). Risk-stratified therapy and dose-dense intensive chemotherapy were adopted in the consolidation therapy. After the second course of therapy, patients in remission were stratified into three risk groups: low-risk children were defined as those with t(8;21) and a white blood cell count lower than 50,000/L, inv(16), or an age younger than 2 years without any high-risk factors; high-risk children were those with CR after consolidation course 1 or induction C , or with abnormalities of monosomy 7, 5q-, t(16;21), t(9;22)(Philadelphia chromosome [Ph1]); intermediate-risk children were those who were not in either a low-risk or high-risk group. Hematopoietic stem cell transplantation (HSCT) was indicated for only relapsed patients in the second CR.
  Interventions: Other: Risk-stratified therapy

INTERVENTIONS:
Other: Risk-stratified therapy — Dose-dense intensive chemotherapy and high dose of Ara-C in the consolidation therapy.
  Groups: CAMS-2009 trial

SUMMARY:
The investigators adopted the CAMS（Chinese Academy of Medical Sciences）-2009 trial for pediatric acute myeloid leukemia (AML) patients between 2009 to 2015, in which a risk-stratified strategy and dose-dense intensive chemotherapy were introduced. The outcomes of CAMS-2009 trial were retrospectively analyzed, and compared to the CAMS-2005 trial.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed AML

Exclusion Criteria:

* children with Down's syndrome and acute promyelocytic leukemia (APL)

Ages: 6 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients admitted to the Department of Pediatrics, Institute of Hematology & Blood Disease Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 320 (Actual)
Dates: Start 2005-04-10 (Actual); Primary Completion 2012-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
overall survival (OS) | From date of diagnosed until the date of death from any cause, assessed up to 60 months
  overall survival
event-free survival (EFS) | From date of diagnosed until the date of first relapse or date of death from any cause, whichever came first, assessed up to 60 months
  event-free survival
complete remission (CR) | through study completion, an average of 1 year
  fewer than 5% blast cells in the bone marrow aspirate and the absence of extramedullary involvement (EMI)

CONTACTS AND LOCATIONS:
Overall Officials: Zhu Xiaofan, Study Chair — Institute of Hematology & Blood Disease Hospital
Locations (1):
- InstituteHBDH, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
The outcomes of CAMS（Chinese Academy of Medical Sciences）-2009 trial are retrospectively analyzed, and compared to the CAMS-2005 trial.